CLINICAL TRIAL: NCT05800171
Title: A Prospective Cohort Study on the Efficacy of Single Use Disposable Elevator Cap (DEC) Duodenoscopy
Brief Title: Efficacy of Single Use Disposable Elevator Cap (DEC) Duodenoscopy
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2301-097-1396
Record Dates: First submitted 2023-03-23; First posted 2023-04-05 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-02

CONDITIONS: Cholangitis
Keywords: Single use disposable elevator cap duodenoscope; Cholangitis
MeSH Terms: conditions — Cholangitis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Weeks
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The goal of this prospective cohort observational study is to compare incidence of cholangitis cause by multi-drug resistant pathogens in patient who underwent ERCP.

The main question it aims to answer are:

* Is the single use disposable elevator cap duodenoscope more effective in preventing cholangitis caused by MDR than fixed cap duodeoscope?
* Is the single use disposable elevator cap duodenoscope more effective in preventing severe cholangitis than fixed cap duodenoscope?

Participants will undergo and ERCP procedure. Among the patients who received the procedure, those who developed cholangitis after procedure will treated with antibiotics after blood culture test. The result of the post procedure cholangitis group's blood culture test and lab data including LFT will be collected. Researches will compare single use disposable elevator cap duodenoscope group and fixed distal cap duodenoscope group to see if there is difference in the incidence of cholangitis caused by MDR pathogens.

DETAILED DESCRIPTION:
Insufficient disinfection of duodenoscopes, particularly the elevator site, can cause ERCP-related infections and serve as a significant source of multidrug-resistant (MDR) infection. To address this issue, a disposable elevator cap (DEC) was developed, and a recent randomized clinical trial demonstrated its effectiveness in reducing contamination following high-level disinfection. However, there is limited evidence in actual clinical practice to reduce cholangitis caused by MDR pathogens. This study aimed to compare the efficacy of the novel DEC duodenoscope with the standard duodenoscope in preventing infection transmission.

We conducted a prospective non-randomized cohort study in a single institution comparing baseline characteristics, technical performance, and incidence of acute cholangitis, including MDR pathogen, in 95 patients using a standard duodenoscope and 101 patients using a DEC duodenoscope.

Age, sex, comorbidities, and indication for ERCP were similar between the two groups. However, the standard duodenoscope group had a higher proportion of naïve papilla (51% vs. 34%, p = 0.04), while the technical success rate was slightly higher in the DEC duodenoscope group (95% vs. 85%, p = 0.15). The rates of procedure-related adverse events were similar between the two groups (16% for DEC vs. 15% for standard). The incidence of post-ERCP cholangitis was also similar (10% for DEC vs. 11% for standard, p = 0.90). The proportion of post-ERCP cholangitis caused by MDR pathogens was similar in the two groups (1% for DEC vs. 2% for standard, p = 0.39).

This study suggests that the technical performance of the DEC duodenoscope is similar to that of the standard duodenoscope. However, more clinical data are needed to confirm the efficacy of the DEC duodenoscope in preventing ERCP-related infection transmission.

ELIGIBILITY:
Inclusion Criteria:

* Patient who undergone ERCP
* 19 years age or older

Exclusion Criteria:

* Patients who already undergone biliary drainage
* Patient who already confirmed of multidrug resistant bacterial infection
* Pregnant women

Min Age: 19 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2023-04-24 (Actual); Primary Completion 2024-02-21 (Estimated); Study Completion 2025-02-21 (Estimated)

PRIMARY OUTCOMES:
Incidence of cholangitis cuased by MDR pathogens | complication with in 2weeks after ERCP
  percentage

CONTACTS AND LOCATIONS:
Overall Officials: Myeong Hwan Lee, M.D, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, Jongno-gu, South Korea